CLINICAL TRIAL: NCT06633445
Title: Evaluation of 3D Guided Botulinum Toxin Type A Injection in Lateral Pterygoid Muscle for Management of Patients With Anterior Disc Displacement With Reduction ( a Randomized Controlled Clinical Trial )
Brief Title: Injecting Lateral Pterygoid Muscle by Botulinum Toxin Type A With 2 Different Methods : 3D Guided Appliance and Electromyography (EMG) .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahmoud Akram Khodir (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Akram Khodir, Assistant Lecturer of oral and maxillofacial surgery, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3D guided Botox injection
Record Dates: First submitted 2024-10-01; First posted 2024-10-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Anterior Disc Displacement
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 3D guided botulinum toxin injection arm (Experimental)
  Interventions: Procedure: botulinum toxin type A injection in lateral pterygoid muscle
- Electromyography botulinum toxin injection arm (Active Comparator)
  Interventions: Procedure: botox injection in lateral pterygoid muscle

INTERVENTIONS:
Procedure: botulinum toxin type A injection in lateral pterygoid muscle — * Needle insertion guide will be placed on upper teeth.
  * Needle will be inserted from needle insertion sleeve and 25-30 units of botulinum toxin type A will be injected.
  * Aspiration will be done before injection, and then, the patient will be asked to manipulate the mandible to activate the lateral pterygoid muscle.
  Arms: 3D guided botulinum toxin injection arm
Procedure: botox injection in lateral pterygoid muscle — * A 27- gauge needle electrode will be inserted lateral to the maxillary tuberosity, just above the maxillary molars to inject 25-30 units of botulinum toxin type A under electromyographic guidance.
  * Aspiration will be done before injection, and then the patient will be asked to manipulate the mandible to activate the lateral pterygoid muscle.
  * The intramuscular injection will be confirmed when the electromyographic device produces a distinct loud sound.
  Arms: Electromyography botulinum toxin injection arm

SUMMARY:
The goal of this study is to evaluate intra-oral botulinum toxin type A injection into lateral pterygoid muscle using a surgical guide synthesized by virtual planning based on CT with soft tissue window.

* To evaluate improvement of maximum interincisal opening (MIO) before and after injection.
* To assess change in disc position before and after injection.
* To evaluate recovery of symptoms as clicking, tenderness of TMJ and tenderness of lateral pterygoid muscle after injection.

Researchers will compare intra-oral botulinum toxin type A injection using a surgical guide synthesized by virtual planning based on CT with soft tissue window to conventional EMG guided botulinum toxin injection into lateral pterygoid muscle in patient with anterior disc displacement with reduction.

Participants will be injected with botulinum toxin type A by intraoral approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes that are diagnosed with ADDWR according to DC/TMD.
2. Their age range between 20 and 45 years.
3. Angle class I maxilla-mandibular relation.

Exclusion Criteria:

1. Patients with degenerative joint disease, musculoskeletal, neuromuscular disorders, cardiovascular, bleeding disorders, breathing difficulties, neurological disorders.
2. Pregnancy and lactating women.
3. History of surgical TMJ intervention.
4. Botox hypersensitivity
5. History of tumors or maxillofacial trauma.
6. Posteriorly edentulous saddles or anterior open bite.
7. Patient contraindicated to MRI examination

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
• Maximum interincisal opening in millimeters. | 6 months
  measured in millimeters from incisal edge of uppercentrals to incisal edge of lower incisors by disposable rulers.
clicking | 6 months
  Any noticeable sound detected temporomandibular joint during opening and closing
temporomandiular joint tenderness | 6 months
  using visual analogue scale to measure pain intensity diagrammed in a line with two ends representing 0 ( no pain) and 10 ( the worst pain) after lateral and auriculotemporal palpation of temporomandibular joint
lateral pterygoid muscle tenderness | 6 months
  using visual analogue scale to measure pain intensity diagrammed in a line with two ends representing 0 ( no pain) and 10 ( the worst pain) after intraoral palpation of lateral pterygoid muscle behind tuberosity

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Raafa N, Melek L, Zoheir H, Mansour E, Sakr A. A novel fully guided technique for botulinum toxin injection in lateral pterygoid muscle using muscle segmentation for TMJ disc displacement with reduction: a randomized controlled trial. BMC Oral Health. 2025 Jun 21;25(1):957. doi: 10.1186/s12903-025-06372-w. PMID 40544291